CLINICAL TRIAL: NCT05555186
Title: Effect of School Based Ambient Bright White Light Intervention on Adolescents´ Sleep Quality, Depression and Mood
Brief Title: The Effects of Bright Light Therapy on Adolescent's Sleep Quality and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reykjavik University (Other)
Collaborators: The Icelandic Research Fund (Unknown)
Responsible Party: Principal Investigator, Birna Baldursdottir, Lecturer, Reykjavik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSN-21-143; 217543-051 (Other Grant/Funding Number: The Icelandic Research Fund)
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disturbance; Depression; Mood; Circadian Rhythms
Keywords: Light Therapy; Sleep Disturbance; Adolescents; Well-being; Circadian Rhythms
MeSH Terms: conditions — Parasomnias; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental light: Sleep quality and well-being (Experimental): Exposure to experimental systematic light exposure (BWL) in classroom where students are located every school day from 8:30 AM until the school finishes between 3 and 4 PM
  Interventions: Device: BWL classrooms (Experimental)
- Comparison light: Sleep quality and well-being (Sham Comparator): Exposure to comparison systematic light exposure (DWL) in classroom where students are located every school day from 8:30 AM until the school finishes between 3 and 4 PM
  Interventions: Device: DWL classrooms (Comparison)
- Unchanged lightning (No Intervention): Conventional lightning in classrooms where students are located every school day from 8:30 AM until the school finishes between 3 and 4 PM

INTERVENTIONS:
Device: BWL classrooms (Experimental) — Adolescents in the BWL classrooms will be exposed to the circadian stimulating bright light (600-1000lx) to maintain alertness. The programming of the LED lighting system in the intervention group (BWL) will be tuned to provide equal stimuli to the cone and melanopsin-containing photoreceptors measured at the eye height (1.2 m above floor level for sitting position) approximately in the range 4500 -5500 K (cool white light) or between 600 and 1000 lx.
  Arms: Experimental light: Sleep quality and well-being
Device: DWL classrooms (Comparison) — Participants in DWL classrooms will receive conventional light from the same kind of equipment as used for the intervention group, only not applying high circadian stimulation(300lx). In order to replicate conventional lighting in the classrooms, the programming of the new LED lighting system in the control group (DWL) will meet the minimum requirements according to EN12464-181, or at least 300 lx measured at table height for a light source rated at 3000 K (warm white light).
  Arms: Comparison light: Sleep quality and well-being

SUMMARY:
Sleep problems are common among adolescents which can have a variety of serious biological, emotional, cognitive and psychological consequences. Numerous studies have shown that adolescents who suffer from insufficient sleep and poor sleep quality experience decreased mental well-being which is a growing concern in modern societies.

Effective interventions that enhance sleep quality among adolescents are lacking. One possible reason for sleep problems among adolescents is disturbance in the body's circadian rhythms. As light is known to be the main coordinating factor in circadian rhythms, light therapy is an auspicious method which aims to entrain the circadian rhythms, thereby enhancing sleep quality and well-being. Indeed, bright light therapy (BLT) has been shown to be a promising treatment to improve sleep and decrease depressive symptoms among different patient groups. However, BLT interventions among healthy adolescents are needed. Therefore, the current study will investigate whether BLT in classrooms of 16 year old students can improve their sleep quality and well-being. The results from the study can be important as it is the first one to examine whether light intensity in the classroom affects sleep and well-being among adolescents. Furthermore, if the hypothesis will be supported, a simple and relatively inexpensive method can be implemented to promote better sleep quality and thus have an extensive effect on adolescents' well-being.

Aim 1 - Assess whether BLT will improve sleep quality of adolescents. Aim 2 - Assess whether BLT will decrease depressive symptoms in adolescents. Aim 3 - Assess whether BLT will improve mood in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* First-year students at the school where the research takes place.
* Participants provide written informed consent.
* Parents or caregivers of participants provide informed consent.
* Read and write Icelandic.

Exclusion Criteria:

* Not first-year students.
* Participant or parent does not provide written informed consent.
* Not capable of reading and writing Icelandic.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
ActTrust: Sleep/wake activity | Up to 9 months
  Measure of night-time and daytime sleep (combined minutes of sleep, sleep-onset latency, and sleep efficiency. Recorded by a wrist actigraph (ActTrust).
ActTrust: Circadian Activity Rhythms | Up to 9 months
  Rest-activity patterns (amplitude, acrophase, mesor) recorded by a wrist actigraph (ActTrust), combined into a circadian activity variable.
ActTrust: Daily physical activity | Up to 9 months
  Measure recorded by a wrist actigraph (ActTrust) showing activity levels of participants.
ActTrust: Environmental light exposure | Up to 9 months
  Measure recorded by a wrist actigraph (ActTrust), showing the types of light a participant is exposed to.
Pittsburgh Sleep Quality Index | Up to 9 months
  The Pittsburgh Sleep Quality Index assesses sleep quality. his measure is composed of 19 items that generate seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). The sum of the seven component scores yields one global score. A person with a global score above 5 is considered to have sleep disturbances. The scale has the test-retest reliability of r=.85 and estimated internal consistency of α=.80.
The Warwick-Edinburgh Mental Well-being Scale | Up to 9 months
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS), 7 item short version will be used to assess overall well-being during the last two weeks. Each item on the list is rated on a 5-point Likert scale ranging from "never" to "very often".
Munich Chronotype Questionnaire (MCTQ) | Up to 9 months
  The Munich Chronotype Questionnaire (MCTQ) is a self-reported measure of chronotype that addresses questions related to sleep and wakefulness. The participants were asked to answer the list based on experience of a typical week in their current situation.
PROMIS cognitive function and cognitive abilities 8a | Up to 9 months
  PROMIS® (Patient-Reported Outcomes Measurement Information System) cognitive function and cognitive abilities 8a consist of 8 self-report item rated on a five point Likert scale ranging from "never" to "very often" on the Cognitive Function scale and "not at all" to "very much" on the Cognitive Abilities scale. Both PROMIS item banks show good psychometric properties, such as a high internal consistency (α =.94 for each).
Depression Anxiety Stress Scales (DASS 21) | Up to 9 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The participants were asked to read the following statement and circle a number 0, 1, 2 or 3 which indicates how much the statement applied to the participant over the past week.
The Cleveland Adolescent Sleepiness Questionnaire | Up to 9 months
  The Cleveland Adolescent Sleepiness Questionnaire (CASQ), a brief, self-completed instrument to measure excessive daytime sleepiness in adolescents. For each statement, the participants were asked to mark the circle under the response that best fits with how often it applies to them. Each item on the list is rated on a 5-point Likert scale ranging from "never" to "almost daily".
Adolescents Daytime Naps | Up to 9 months
  Adolescents Daytime Naps measure how often participants fall asleep daily. If they rest or fall asleep during the day, it is called a day-nap, whether they have planned to go to bed or not. Daytime hours also cover shorter periods of time when they rest or fall asleep, for example over a computer / television or reading. First participants are asked about daytime hours on weekdays and then about daytime hours on weekends. If participants go to bed more than once a day, they should record the total time staying in bed.
Adolescents Screen Time | Up to 9 months
  The participants were asked how long time they spend on a computer, tablet, game console, television, phone or other display device in the following: school lessons, work/internship, computers or social media. The answer possibilities are 0-23 hours and 0-50 minutes.
Physical activity | Up to 9 months
  The participants were asked two questions about their physical activity during the last seven days. The participants were asked how long time per one day they usually spend participating in physical activity. Include the time they spent waking, jogging, running, cycling, exercising or doing some kind of sport. The answer possibilities range from "less than 1/2 hour a day" up to "more than 6 hours a day" The participants were also asked how many days of the last seven days they participated in physical activity for at least 60 minutes so that their heart rate increased and they sometimes got out of breath. The participation may include physical activity, workout, brisk walking, cycling in free time or transportation between different locations. The answers range from "almost never" up to "seven days".
Sedentary behaviour | Up to 9 months
  The participants were asked how long time they usually spend sitting the last seven days. The period starts when they wake up in the morning and ends when they goes to bed for the night. Include time spent at work, at school, at home, and in their free time. This can include time spent at a desk, dining table, visiting, watching movies, reading, or in front of a television, computer, or other monitor. The answer possibilities range from "30 minutes per day" up to "more than 16 hours per day".

CONTACTS AND LOCATIONS:
Overall Officials: Birna Baldursdottir, PhD, Principal Investigator — Reykjavik University; Heiddis B. Valdimarsdottir, PhD, Study Chair — Reykjavik University
Locations (1):
- Reykjavik University, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger AT, Wahlstrom KL, Widome R. Relationships between sleep duration and adolescent depression: a conceptual replication. Sleep Health. 2019 Apr;5(2):175-179. doi: 10.1016/j.sleh.2018.12.003. Epub 2019 Jan 30. PMID 30928118
- [Background] Brand S, Lemola S, Mikoteit T, Holsboer-Trachsler E, Kalak N, Bahmani DS, Puhse U, Ludyga S, Gerber M. [Sleep and Psychological Functioning of Children and Adolescents - a Narrative Review]. Prax Kinderpsychol Kinderpsychiatr. 2019 Feb;68(2):128-145. doi: 10.13109/prkk.2019.68.2.128. German. PMID 30757973
- [Background] Chaput JP, Gray CE, Poitras VJ, Carson V, Gruber R, Olds T, Weiss SK, Connor Gorber S, Kho ME, Sampson M, Belanger K, Eryuzlu S, Callender L, Tremblay MS. Systematic review of the relationships between sleep duration and health indicators in school-aged children and youth. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S266-82. doi: 10.1139/apnm-2015-0627. PMID 27306433
- [Background] Chang AM, Aeschbach D, Duffy JF, Czeisler CA. Evening use of light-emitting eReaders negatively affects sleep, circadian timing, and next-morning alertness. Proc Natl Acad Sci U S A. 2015 Jan 27;112(4):1232-7. doi: 10.1073/pnas.1418490112. Epub 2014 Dec 22. PMID 25535358
- [Background] Gariepy G, Danna S, Gobina I, Rasmussen M, Gaspar de Matos M, Tynjala J, Janssen I PhD, Kalman M PhD, Villerusa A, Husarova D, Brooks F, Elgar FJ, Klavina-Makrecka S MSc, Smigelskas K, Gaspar T, Schnohr C. How Are Adolescents Sleeping? Adolescent Sleep Patterns and Sociodemographic Differences in 24 European and North American Countries. J Adolesc Health. 2020 Jun;66(6S):S81-S88. doi: 10.1016/j.jadohealth.2020.03.013. PMID 32446613
- [Background] Gradisar M, Gardner G, Dohnt H. Recent worldwide sleep patterns and problems during adolescence: a review and meta-analysis of age, region, and sleep. Sleep Med. 2011 Feb;12(2):110-8. doi: 10.1016/j.sleep.2010.11.008. Epub 2011 Jan 22. PMID 21257344